CLINICAL TRIAL: NCT05439720
Title: Acute Effect of Exogenous Ketosis on Sleep Architecture Following Morning and Evening Strenuous Exercise
Brief Title: Acute Effect of Exogenous Ketosis on Sleep Architecture Following Strenuous Exercise
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Peter Hespel, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: S65394
Record Dates: First submitted 2022-06-16; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Sleep
Keywords: Ketone; Exercise; Sleep
MeSH Terms: conditions — Ketosis; Motor Activity | interventions — formic acid 4-(3-oxobutyl)phenyl ester; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Exercise and ketone (Experimental): Ketone ester is provided
  Interventions: Dietary Supplement: Ketone ester; Behavioral: Exercise
- Exercise and placebo (Placebo Comparator): Placebo is provided
  Interventions: Dietary Supplement: Placebo; Behavioral: Exercise
- Non-exercise and placebo (Placebo Comparator): Placebo is provided
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone ester — A dose of 25g of ketone ester after each training session and 30 minutes before sleeptime. The total dose is 75g of ketone ester.
  Arms: Exercise and ketone
Dietary Supplement: Placebo — Collagen peptan (3g) mixed with 1 mM bitter sucrose octaacetate and 20ml of pure water. A dose of 25g of placebo drink is provided after each training session and 30 minutes before sleeptime. The total dose is 75g of placebo drink.
  Arms: Exercise and placebo; Non-exercise and placebo
Behavioral: Exercise — A 120 minutes cycling endurance training session (ET) two hours after breakfast and an evening high-intensity-interval training (HIIT) ending one hour before bedtime
  Arms: Exercise and ketone; Exercise and placebo

SUMMARY:
The aim of this study is to investigate the effect of oral ketone ester administration on sleep architecture. To investigate this, the investigators use a randomised, placebo-controlled, cross-over research design. The study comprises three experimental sessions, each separated by a one-week washout period. Two of the three experimental sessions consist of a 120 minutes cycling endurance training session (ET) two hours after breakfast and an evening high-intensity-interval training (HIIT) ending one hour before bedtime. After each training session, and 30 minutes before sleeptime, subjects receive a ketone ester or a control drink . To investigate the effects of strenuous exercise on sleep alone, an additional experimental session without exercise is added.

Before bedtime, a venous blood sample is taken to evaluate hormones playing an important role in sleep regulation. During the experimental sessions, the subjects sleep in a sleep facility to evaluate quality of sleep. Time spent in different sleep phases is measured via polysomnography (PSG). Urine output throughout the day and night will be collected for measurement of urinary excretion of adrenaline and noradrenaline as an index of intrinsic sympathetic activity.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 and 35 years old
* Recreational or competitive cyclists performing regularly cycling training sessions with an average training volume of more than 6 hours per week
* Good health status confirmed by a medical screening
* Body Mass Index (BMI) between 18 and 25
* Normal sleep pattern as assessed by the Pittsburgh Sleep Quality Index (PSQI)
* Moderate sleep chronotype, assessed by the Horne and Östberg questionnaire

Exclusion Criteria:

* Excessive daytime sleepiness as assessed by the Epworth scale
* Depression or anxiety as assessed by the Beck Depression Inventory and Beck Anxiety Inventory
* Night-shifts or travel across time zones in the month preceding the study
* Any kind of injury/pathology that is a contra-indication to perform high-intensity exercise
* Intake of any medication or nutritional supplement that is known to affect exercise performance or sleep
* Smoking
* Involvement in elite athletic training at a semi-professional or professional level
* Current participation in another research trial
* Any other argument to believe that the subject is unlikely to successfully complete the full study protocol

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Total sleep time | Between each condition, interspersed each time with a one-week wash-out period (The total duration of the measurements is two weeks)
  Change in total sleep time between conditions as evaluated with polysomnography
Urinary nocturnal adrenaline excretion | Between each condition, interspersed each time with a one-week wash-out period (The total duration of the measurements is two weeks)
  Change in urinary nocturnal adrenaline excretion between conditions
Urinary nocturnal noradrenaline excretion | Between each condition, interspersed each time with a one-week wash-out period (The total duration of the measurements is two weeks)
  Change in urinary nocturnal adrenaline excretion between conditions

SECONDARY OUTCOMES:
Total rapid-eye-movement sleep | Between each condition, interspersed each time with a one-week wash-out period (The total duration of the measurements is two weeks)
  Change in total rapid-eye-movement sleep between conditions as evaluated with polysomnography
Total non-rapid-eye-movement sleep | Between each condition, interspersed each time with a one-week wash-out period (The total duration of the measurements is two weeks)
  Change in total non-rapid-eye-movement sleep between conditions as evaluated with polysomnography
Total slow-wave sleep | Between each condition, interspersed each time with a one-week wash-out period (The total duration of the measurements is two weeks)
  Change in total slow-wave sleep between conditions as evaluated with polysomnography
Plasma adrenaline concentration | Between each condition, interspersed each time with a one-week wash-out period (The total duration of the measurements is two weeks)
  Change in plasma adrenaline concentration between conditions
Plasma noradrenaline concentration | Between each condition, interspersed each time with a one-week wash-out period (The total duration of the measurements is two weeks)
  Change in plasma noradrenaline concentration between conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Physiology Group, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Robberechts R, Albouy G, Hespel P, Poffe C. Exogenous Ketosis Improves Sleep Efficiency and Counteracts the Decline in REM Sleep after Strenuous Exercise. Med Sci Sports Exerc. 2023 Nov 1;55(11):2064-2074. doi: 10.1249/MSS.0000000000003231. Epub 2023 Jun 1. PMID 37259248